CLINICAL TRIAL: NCT02783079
Title: Insomnia Interventions in Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-146EX
Record Dates: First submitted 2016-02-12; First posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Insomnia
Keywords: Breast Cancer; Prostate Cancer; Colon Cancer; Lung Cancer; Gynecologic Cancer
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Lung Neoplasms | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Cognitive Behavioral Therapy (CBT)
  Interventions: Behavioral: CBT
- Arm 2 (Active Comparator): Mindfulness Based Stress Reduction (MBSR)
  Interventions: Behavioral: MBSR

INTERVENTIONS:
Behavioral: CBT
  Other Names: cognitive behavioral therapy
  Arms: Arm 1
Behavioral: MBSR
  Other Names: mindfulness based stress reduction
  Arms: Arm 2

SUMMARY:
This study looks at two different interventions used for the treatment of insomnia in survivors of breast, colon, lung, prostate and gynecologic cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate two validated interventions for the treatment of insomnia in cancer survivors of breast, colon, lung and prostate cancer. Moreover, it will provide an opportunity to assess the efficacy of both of these interventions in a group setting in patients of varied ethnic backgrounds including African-Americans, Latinos and Caucasians. The results of this study will help clinicians provide future interventions specific to cancer type and ethnicity in order to better serve the needs of our cancer survivors and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age 18 and over
* diagnosis of breast, colon, lung, prostate or gynecologic cancer that is non metastatic
* receiving treatment at one of the outpatient offices of the MD Anderson Cancer Center at Cooper
* Self reported insomnia
* Not currently taking any medications to treat insomnia
* No medical or psychological condition that would prevent successful protocol completion in the opinion of investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Baseline to 6 weeks and 6 weeks to 12 weeks
  Change in Insomnia Severity Index (ISI) rating ratings in cancer survivors receiving CBT vs. MBSR interventions.

SECONDARY OUTCOMES:
Change in Brief Fatigue Inventory (BFI) | Baseline to 6 weeks and 6 weeks to 12 weeks
  Change in Fatigue rating using the BFI in cancer survivors receiving CBT vs. MBSR interventions.
Change in Depression, Anxiety and Stress Scale 21 (DASS21) | Baseline to 6 weeks and 6 weeks to 12 weeks
  Change in Depression and Anxiety rating using the DASS21 in cancer survivors receiving CBT vs. MBSR interventions
Number of patients who respond to CBT vs MBSR based on Ethnicity | 12 weeks
  Variations in efficacy outcomes based on ethnicity

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - MD Anderson Cancer Center at Cooper, Voorhees Township, New Jersey